CLINICAL TRIAL: NCT05084235
Title: Empagliflozin to Elderly and Obese Patients With Cardiovascular Disease (Empire Prevent: Cardiac): A Randomized Controlled Trial
Brief Title: The Cardiac Effects of Empagliflozin in Patients With High Risk of Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jacob Moller (Other)
Collaborators: Danish Heart Foundation (Other); Herlev and Gentofte Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Hillerod Hospital, Denmark (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jacob Moller, Professor, MD, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-20210028-1
Record Dates: First submitted 2021-09-03; First posted 2021-10-19 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; Obesity
MeSH Terms: conditions — Heart Failure; Obesity | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empaglifloxin (Active Comparator)
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Patients are randomized 1:1 to receive either Empagliflozin or matching placebo for 180 days
  Arms: Empaglifloxin
Drug: Placebo — Placebo matches the active drug in appearance, odor and labelling
  Arms: Placebo

SUMMARY:
The aim of this trial is to assess the effect of Empagliflozin on cardiac mass, volumes, cardiac biomarkers, metabolism, daily activity level, health-related quality of life in patients in elderly and obese patients with increased risk of developing heart failure. The primary hypotheses are that 180 days of treatment with Empagliflozin 10 mg a day will: 1) reduce left ventricular mass index, and 2) increase peak VO2 (maximal oxygen consumption) compared with placebo.

DETAILED DESCRIPTION:
The Empire Prevent: Cardiac is a part of the Empire Prevent Trial Program, which also comprises the Empire Prevent: Metabolic

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >28kg/m2
* Age 60-84 years
* Established risk factor for developing heart failure, defined as at least one of the following:
* hypertension
* ischemic heart disease
* stroke/transient cerebral ischemia
* chronic kidney disease (eGFR 30-45ml/min/1.73m2)

Exclusion Criteria:

* Diabetes mellitus type 1 or 2 (no medical history, no antidiabetic treatment)
* Heart failure with reduced ejection fraction (LVEF <40%)
* Inability to perform exercise test
* Dementia
* Severe non-compliance
* Substance abuse
* Severe chronic obstructive pulmonary disease (FEV1<50% expected value)
* Permanent atrial fibrillation
* GFR <30 ml/min/1,73m2
* Severe peripheral artery disease
* Cancer treatment within one year beside prostate cancer and basal cell carcinoma
* Severe aortic or mitral valve disease
* Pregnancy or breastfeeding
* Acute hospital admission within 30 days
* Participation in other pharmacological study

Ages: 60 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass index | 180 days
  Between-group difference in the change of left ventricular mass index (LVMI) assessed by cardiac magnetic resonance image
Maximal oxygen consumption | 180 days
  Between-group difference in the change of maximal oxygen consumption (peak VO2) assessed by cardiopulmonary exercise test

SECONDARY OUTCOMES:
Left ventricular volume | 180 days
  Between-group difference in the change of left ventricular end-diastolic volume index (LVEDVI) and left ventricular end-systolic volume index (LVESVI) assessed by cardiac magnetic resonance image
Left ventricular function | 180 days
  Between-group difference in the change of first phase ejection fraction and left ventricular ejection fraction (LVEF) assessed by cardiac magnetic resonance image
Daily activity level | 180 days
  Between-group difference in the change of daily activity level assessed by accelerometer

OTHER OUTCOMES:
Quality-of-life scores | 180 days
  Between-group difference in the change of self-reported quality of life assessed by the 36-item short form health survey (SF-36 questionnaire). The SF-36 targets eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each item is scored on a scale from 0 to 100, with a higher score representing a more favorable health state. An average score is calculated for each health concept.
Blood pressure | 180 days
  Between-group difference in the change of systolic and diastolic blood pressure assessed by ambulatory blood pressure measurement
Wall stress | 180 days
  Between-group difference in the change of estimated end-systolic wall stress (ESWS). ESWS will be calculated from results of multimodality imaging combining MRI and echocardiography by using a formula incorporating MRI LV end-systolic diameter and wall thickness as well as echocardiographic mean and arterial blood pressure as proposed by Reichek et al. based on the Law of Laplace. (please see references Reichek et al and Carter-Storch et al. in the reference list)
Left atrium size | 180 days
  Between-group difference in the change of left atrial maximal and minimal size measured by cardiac magnetic resonance image
Global strain | 180 days
  Between-group difference in the change of global strain assessed by cardiac magnetic resonance image
Growth differentiation factor 15 | 180 days
  Between-group difference in the change of the biomarker growth differentiation factor 15 (pg/ml)
Cardiac fibrosis | 180 days
  Between-group difference in the change of cardiac fibrosis assessed by cardiac magnetic resonance image
Left atrium function | 180
  Between-group difference in the change of left atrial emptying fraction and left atrium ejection fraction assessed by cardiac magnetic resonance image
Biomarkers of heart disease | 180 days
  Between-group difference in the change of biomarkers of heart disease, including atrial natriuretic peptide (ANP), brain (B-type) natriuretic peptide (BNP), and N-terminal pro-hormone BNP (NT-proBNP). All measured as pmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Eifer Møller, MD, PhD,, Principal Investigator — Odense University Hospital; Morten Schou, MD, PhD, DmSc, Principal Investigator — Herlev-Gentofte Hospital
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reichek N, Wilson J, St John Sutton M, Plappert TA, Goldberg S, Hirshfeld JW. Noninvasive determination of left ventricular end-systolic stress: validation of the method and initial application. Circulation. 1982 Jan;65(1):99-108. doi: 10.1161/01.cir.65.1.99. No abstract available. PMID 7053293
- [Background] Carter-Storch R, Moller JE, Christensen NL, Rasmussen LM, Pecini R, Sondergard E, Videbaek LM, Dahl JS. End-systolic wall stress in aortic stenosis: comparing symptomatic and asymptomatic patients. Open Heart. 2019 Apr 9;6(1):e001021. doi: 10.1136/openhrt-2019-001021. eCollection 2019. PMID 31168387
- [Derived] Andersen CF, Larsen JH, Jensen J, Omar M, Nouhravesh N, Kistorp C, Tuxen C, Gustafsson F, Knop FK, Forman JL, Davidovski FS, Jensen LT, Hojlund K, Kober L, Antonsen L, Poulsen MK, Schou M, Moller JE. Empagliflozin to elderly and obese patients with increased risk of developing heart failure: Study protocol for the Empire Prevent trial program. Am Heart J. 2024 May;271:84-96. doi: 10.1016/j.ahj.2024.02.005. Epub 2024 Feb 15. PMID 38365073

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT05084235/SAP_000.pdf